CLINICAL TRIAL: NCT04218279
Title: The EMS Sleep Health and Fatigue Study: A Randomized Controlled Trial
Brief Title: The EMS Sleep Health Study: A Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial enrollment terminated early due to end of funding period.
Sponsor: University of Pittsburgh (Other)
Collaborators: National Highway Traffic Safety Administration (NHTSA) (U.S. Federal Agency); National Association of State EMS Officials (Other)
Responsible Party: Principal Investigator, Daniel Patterson, PhD, NRP, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY19080090; DTNH2215R00029 (Other Grant/Funding Number: National Highway Traffic Safety Administration (NHTSA))
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Sleep Quality; Fatigue
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Masking Description: Unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Health Education (Experimental): At baseline, the experimental group will have immediate access to 10 brief education modules focused on diverse elements of sleep health and fatigue.
  Interventions: Other: Sleep Health Education
- Wait List Control (Active Comparator): At 3 months after baseline, the wait-list control group will be provided access to the 10 education modules focused on diverse elements of sleep health and fatigue..
  Interventions: Other: Sleep Health Education

INTERVENTIONS:
Other: Sleep Health Education — Intervention materials include 10 brief education modules that the target population will review/view on a secure study-specific website.

SUMMARY:
The experiment seeks to determine the impact of a sleep health and fatigue education and training program on diverse indicators of sleep and fatigue among Emergency Medical Services (EMS) personnel. The overarching goals of this research study are to [1] enhance our understanding of the relationships between shift work, sleep, and fatigue in EMS operations; and [2] determine whether or not providing education and training to EMS personnel on the importance of sleep health and dangers of fatigue impact indicators of sleep and fatigue. The investigators will accomplish these goals by using a cluster-randomized trial study design with a wait-list control group.

DETAILED DESCRIPTION:
The overarching goals of this research study are to:

1. enhance our understanding of the relationships between shift work, sleep, and fatigue in EMS operations; and
2. determine whether or not providing education and training to EMS personnel on the importance of sleep health and dangers of fatigue impact indicators of sleep and fatigue.

The investigators will recruit EMS nationwide for EMS agencies to participate in this study and focus on moderately sized EMS agencies with between 50 and 300 employees (yet we will not outright exclude smaller or larger organizations). Agencies that run dual ground-based and air-medical EMS services are eligible. Maximum enrollment at the agency-level is n=30 EMS agencies. Agencies will be randomized upon enrollment to one of two arms: [1] Intervention group; or [2] the Wait-List control group. The intervention group will receive immediate access to the intervention materials (the 10 brief Sleep Health Education Modules). The wait-list control group will receive access to intervention materials at 3 months post enrollment/baseline.

Within each agency, the investigators will recruit individual EMS clinicians to participate. Goal enrollment within each agency is a minimum of 30 and a maximum of 50 EMS clinicians.

All individual EMS clinician participants will undergo informed consent, answer a baseline survey, and be queried via mobile phone text message at regular intervals which will begin upon enrollment. These mobile phone text message queries will assess indicators of sleep and fatigue. All participants will be asked to answer two follow up surveys at 3 months and 6 months. The total duration of study participation is 6 months. The primary outcome of interest is sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI). The secondary outcome of interest is fatigue as measured by the Chalder Fatigue Questionnaire (CFQ).

ELIGIBILITY:
Inclusion Criteria:

* EMS Personnel:

  1. 18 years of age or older
  2. Currently working as an EMS clinician
  3. Working a minimum of one shift a week
  4. Working & residing in the United States
  5. Working at one of the EMS organizations that agreed to participate in this study
  6. Have a cellular, mobile, or smart phone that can send and receive text messages
  7. Willing to answer online surveys and respond to text-message queries for seven days in a row every third week of the month for a total of 24 weeks/6 months

Exclusion Criteria:

* EMS Personnel:

  1. Individuals <18 years of age
  2. Not currently working as an EMS clinician
  3. Does not work a minimum of one shift a week
  4. Does not work and/reside in the United States
  5. Does not work at one of the EMS organizations that agreed to participate in this study
  6. Does not have a cellular, mobile, or smart phone that can send and receive text messages
  7. Is not willing to answer online surveys and respond to text-message queries for seven days in a row every third week of the month for a total of 24 weeks/6 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Patterson, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual de-identified participant data collected during the trial will be shared with the funding organization (the National Highway Traffic Safety Administration (NHTSA)) and with researchers who provide a methodologically sound proposal and have been approved by the funding organization and by the University of Pittsburgh.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified data will be made available immediately following publication and upon approval from the funding organization. No end date.
Access Criteria: Access will be provided to researchers who provide a methodologically sound proposal and have been approved by the funding organization and by the University of Pittsburgh.

REFERENCES:
- [Derived] Patterson PD, Martin SE, MacAllister SA, Weaver MD, Patterson CG. Variations in Sleep, Fatigue, and Difficulty with Concentration Among Emergency Medical Services Clinicians During Shifts of Different Durations. Int J Environ Res Public Health. 2025 Apr 6;22(4):573. doi: 10.3390/ijerph22040573. PMID 40283798
- [Derived] Patterson PD, Martin SE, Brassil BN, Hsiao WH, Weaver MD, Okerman TS, Seitz SN, Patterson CG, Robinson K. The Emergency Medical Services Sleep Health Study: A cluster-randomized trial. Sleep Health. 2023 Feb;9(1):64-76. doi: 10.1016/j.sleh.2022.09.013. Epub 2022 Nov 10. PMID 36372657

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: EMS Agencies
Period: Overall Study
Arm/Group | Sleep Health Education | Wait List Control
Started | 316; 16 EMS Agencies | 362; 20 EMS Agencies
Completed | 211; 15 EMS Agencies | 225; 20 EMS Agencies
Not Completed | 105; 1 EMS Agencies | 137; 0 EMS Agencies

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Health Education | Wait List Control | Total
Number analyzed (Participants) | 316 | 362 | 678
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (9.6) | 37.4 (10.1) | 38.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Some participants did not answer the question about sex.
  Participants
    number analyzed (Participants) | 302 | 347 | 649
    Female | 97 | 92 | 189
    Male | 205 | 255 | 460
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Some participants did not complete the survey.
  Participants
    number analyzed (Participants) | 302 | 348 | 650
    Hispanic or Latino | 16 | 18 | 34
    Not Hispanic or Latino | 274 | 322 | 596
    Unknown or Not Reported | 12 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Some participants did not complete the survey.
  Participants
    number analyzed (Participants) | 302 | 348 | 650
    American Indian or Alaska Native | 3 | 7 | 10
    Asian | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 4 | 5
    White | 284 | 320 | 604
    More than one race | 8 | 8 | 16
    Unknown or Not Reported | 6 | 7 | 13
Mean Pittsburgh Sleep Quality Index Score [Mean (Standard Deviation); unit: units on a scale] — Minimum score possible = 0. Maximum score possible = 21. Higher is worse indicating poorer sleep quality.
  units on a scale | 8.77 (3.3) | 8.96 (3.6) | 8.87 (3.5)
Mean Chadler Fatigue Questionnaire Score [Mean (Standard Deviation); unit: units on a scale] — Minimum score possible = 0. Maximum score possible = 11. Higher score indicating worse mental and physical fatigue. Population: Some participants did not complete the survey.
  units on a scale
    number analyzed (Participants) | 302 | 348 | 650
    (all) | 6.64 (2.6) | 6.55 (2.8) | 6.6 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sleep Quality at 3 Months
Description: Sleep quality will be measured with the Pittsburgh Sleep Quality Index (PSQI) tool. Scores range from 0-21 with scores greater than or equal to 6 classified as poor sleep quality.
Time Frame: baseline to 3 months
Population: Complete cases
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sleep Health Education | Wait List Control
Number analyzed (Participants) | 209 | 223
units on a scale | -0.53 (2.64) | -0.08 (2.60)

2. Secondary Outcome: Change From Baseline in Fatigue at 3 Months
Description: Fatigue will be measured with the Chalder Fatigue Questionnaire (CFQ). The CFQ is a brief 11-item survey tool that measures mental and physical fatigue with scores ranging from 0-11. Scores 4 or greater indicate severe fatigue.
Time Frame: baseline to 3 months
Population: Complete cases
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sleep Health Education | Wait List Control
Number analyzed (Participants) | 208 | 222
units on a scale | 0.19 (2.23) | 0.01 (2.45)

ADVERSE EVENTS:
Description: We did not assess for adverse events in this study given the minimal risk and study design.
Arm/Group | Sleep Health Education | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT04218279/Prot_SAP_001.pdf
  • Informed Consent Form (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT04218279/ICF_002.pdf